CLINICAL TRIAL: NCT05953038
Title: Lysergic Acid Diethylamide Occupancy of the Serotonin 2A Receptor in the Human Brain
Brief Title: LSD Occupancy of the Serotonin 2A Receptor in the Human Brain
Acronym: dOccLS
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Gitte Moos Knudsen, Professor, DMsc, MD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-21060056; 2021-002633-42 (EudraCT Number)
Record Dates: First submitted 2023-02-14; First posted 2023-07-19 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Basic Science
Keywords: Lysergic acid diethylamide; PET; Psychedelic; Hallucinogen; Physiological Effects of Drugs; Psychotropic Drugs; Ergolines; Serotonin; Serotonin Agents; Neurotransmitter Agents; Molecular Mechanisms of Pharmacological Action
MeSH Terms: interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Intervention Model Description: Each participant will be given one of 25, 50, 75, 100, 125, 150, 175 or 200 micrograms of lysergic acid diethylamide (LSD) equivalent as freebase.
Masking Description: Participants will be blinded with respect to dose only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LSD dose-ranging group (Experimental): All participants will receive between 25 and 200 micrograms of lysergic acid diethylamide equivalent as freebase, single blinded with respect to dose. Simultaneous PET/MR imaging will be performed during acute drug effects.
  Interventions: Drug: Lysergic Acid Diethylamide Tartrate

INTERVENTIONS:
Drug: Lysergic Acid Diethylamide Tartrate — D-Lysergic Acid Diethylamide (LSD) D-tartrate as oral drinking solution (water / ethanol 20% m/m)
  Other Names: LSD; d-LSD; LSD-25

SUMMARY:
The investigators wish to quantify the relation between administered dose of lysergic acid diethylamide (LSD), plasma LSD levels, and occupancy at the serotonin 2A receptor (5-HT2AR) using [11C]CIMBI-36 positron emission tomography.

DETAILED DESCRIPTION:
Healthy participants will be administered one of a single dose of lysergic acid diethylamide (LSD) between 25 and 200 micrograms equivalent freebase. They will receive [11C]CIMBI-36 positron emission tomography (PET) scans at baseline and twice following LSD administration during peak and declining drug effects. PET scans will be acquired in a simultaneous PET/Magnetic Resonance Imaging (MRI) scanner which will also collect functional brain imaging data. Venous blood samples will be repeatedly drawn during acute drug effects for quantification of plasma LSD levels. Participants will also repeatedly rate their subjective drug intensity on a scale from 0 to 10 during acute drug effects. Together these data will inform the dose-binding relation of LSD at the serotonin (5-HT) 2A receptor, the primary site of action. This data will also inform the relation between 5-HT2A receptor binding by LSD and the induced subjective effects, as well as the effects on functional brain activity as measured with functional MRI.

ELIGIBILITY:
Inclusion Criteria:

• Healthy individual between 18-75 years old

Exclusion Criteria:

* Current or past history of primary psychiatric illness (The Diagnostic and Statistical Manual of Mental Disorders IV axis-I or World Health Organisation International Classification of Diseases-10 diagnostic classification)
* Current or past history of primary psychiatric illness (The Diagnostic and Statistical Manual of Mental Disorders IV axis-I or World Health Organisation International Classification of Diseases-10 diagnostic classification) in a first degree relative (i.e., parents, siblings)
* Current or past history of neurological disease, significant somatic condition/disease
* Use of medication that could potentially influence results (e.g.., drugs that act on relevant components of the serotonin system or may interfere with metabolism of study drug)
* Non-fluent Danish language skills
* Profound visual or auditory impairments
* Severe learning disability
* Pregnancy on the scan date, verified by a pregnancy test (test omitted if confirmed that individual is post-menopausal)
* Lactation (females)
* Contraindications for magnetic resonance imaging (e.g., pacemaker, claustrophobia, etc.)
* Contraindications for positron emission tomography
* Alcohol or drug abuse
* Allergy to administered compounds
* Participant in research study with >10 millisievert exposure within the past year or significant occupational exposure to radioactive substances
* Abnormal ECG (ECG indicating current or previous heart disease or predisposition to heart disease, e.g., QT prolongation) or use of QT prolonging medication
* Use of psychedelic substance within the preceding six months
* Blood donation up to three months before the study (i.e., more than 500ml of blood)
* Head injury or concussion resulting in loss of consciousness for more than 2 min
* Haemoglobin levels < 7.8 mmol/l for women and 8.4 mmol/l for men
* Ferritin levels outside normal range (12-300 µg/L)
* Body-weight < 50 kg or > 110kg
* body-mass index > 35
* Individual assessment by research staff deeming drug administration unsafe due to ethical or psychological circumstance of the participant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2027-12-18 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma LSD - serotonin 2A receptor (5-HT2AR) occupancy relation | Within 24 hours following drug administration
  Occupancy will be estimated by comparing non-displaceable binding potential (BPND) values using baseline and intervention rescans as calculated using a simplified reference tissue model (SRTM). Occupancy values will be compared to plasma lysergic acid diethylamide (LSD) levels.

SECONDARY OUTCOMES:
Subjective drug intensity - 5-HT2AR occupancy relation | Within 24 hours following drug administration
  Occupancy will be calculated as described above. Subjective drug intensity is collected during positron emission tomography (PET) scans by asking participants.
fMRI network disintegration - 5-HT2AR occupancy relation | Within 24 hours following drug administration
  functional magnetic resonance imaging (fMRI) data will be used to estimate functional-network connectivity using a standard functional brain atlas. Then the relation between decreases in functional network connectivity and 5-HT2AR occupancy will be estimated.
fMRI brain entropy - 5-HT2AR occupancy relation | Within 24 hours following drug administration
  fMRI brain entropy will be estimated by the shannon entropy of dynamic conditional correlation of within and between network connectivity as well as the lempel-ziv complexity of concatenated binarised blood-oxygen level dependent (BOLD) signals across regions. The relation between each of these measures with 5-HT2AR occupancy will be estimated.
Cerebral perfusion - 5-HT2AR occupancy relation | Within 24 hours following drug administration
  Cerebral perfusion will be estimated using arterial spin labelling. The relation between this measure and 5-HT2AR occupancy will be estimated.
Administered LSD dose - 5-HT2AR occupancy relation | Within 24 hours following drug administration
  Administered dose (25 to 200 mcg) will be compared with peak LSD occupancy to determine what doses produce maximal occupancy at the 5-HT2AR.

OTHER OUTCOMES:
Hysteresis effect of 5-HT2AR binding | Within 24 hours following drug administration
  Estimated dose-occupancy curves derived from the first PET scan and second PET scan will be calculated separately to evaluate whether there are differences in estimated plasma level-occupancy relation at different timepoints following LSD administration which may indicate a hysteresis effect due to peripheral LSD metabolism without unbinding of LSD from the 5-HT2A receptor.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte M Knudsen, DMsc, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Neurobiology Research Unit, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lab study homepage — https://nru.dk/index.php/research-menu/ongoing-projects/375-lsd-occupancy-of-the-serotonin-2a-receptor-in-the-human-brain-docls